CLINICAL TRIAL: NCT05503290
Title: A Pilot Study for the Lullaby Project as a Musical Intervention for Pregnant Individuals With Epilepsy
Brief Title: The Lullaby Project as a Musical Intervention for Pregnant Individuals With Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Esther Bui, Assistant Professor, MD FRCPC, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-6199
Record Dates: First submitted 2022-08-13; First posted 2022-08-16 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy; Pregnancy Related
Keywords: Music; Empowerment
MeSH Terms: conditions — Epilepsy; Empowerment

STUDY DESIGN:
Intervention Model Description: This study is a randomized-controlled pilot study where enrolled subjects (primiparous individuals with epilepsy) will be randomized 1:1 to the control or intervention group (participation in the Lullaby Project). Outcomes of interest will be measured in each participant at day of consent, 3 weeks after, 7 weeks after, and 10 weeks after. A follow-up via email will be conducted for intervention participants 6 months after their last workshop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Lullaby Project (Active Comparator): Participants assigned to the intervention group will meet virtually with a professional musician for 5-7 sessions over the course of 10 weeks. Each session will last approximately 1.5 hours and will be conducted via Zoom.
  Interventions: Behavioral: Lullaby Project

INTERVENTIONS:
Behavioral: Lullaby Project — Our proposed intervention is the randomized participation of pregnant individuals with epilepsy in the Lullaby Project coordinated by a musical institution in Toronto. The Lullaby Project is an initiative first created by Carnegie Hall's Weill Music Institute. In this program, pregnant women and/or new mothers are paired with professional musicians to compose and write personal lullabies for their child(ren). Since its inception in 2011, the project has expanded globally and have helped numerous families write original lullabies for their newborns. The Lullaby intervention is unlike traditional music therapy as patients are actively participating in the creative song-writing process, not singularly in passive listening. Through sessions, participants will be given an opportunity to share experiences, experiment with musical arrangements, write lyrics, and receive positive feedback from the musician.
  Arms: Lullaby Project

SUMMARY:
This study's proposed intervention is the randomized participation of pregnant individuals with epilepsy in the Lullaby Project coordinated by a musical institution in Toronto. The purpose of this present study is to investigate the potential benefits of the Lullaby Project on pregnant individuals with epilepsy. Namely, effects on quality of life-related to epilepsy, symptoms of depression and anxiety, perceived stress, and feelings of empowerment.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* currently pregnant and primiparous
* able to provide informed consent
* able to have internet access
* have a confirmed diagnosis of epilepsy based on EEG or clinical evidence

Exclusion Criteria:

* need of a language interpreter to provide informed consent and/or communicate with the MH-RTH musician
* prior involvement in the Lullaby Project

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Epilepsy | 6 months
  Assess quality of life related to epilepsy (via QOLIE-31-P, the Patient-Weighted Quality of Life in Epilepsy inventory); minimum value is 0 and maximum value is 100. Higher scores represent better quality of life.

SECONDARY OUTCOMES:
Depression and Anxiety | 6 months
  Assess symptoms of depression and anxiety (via DASS-21, the Depression, Anxiety and Stress Scale - 21 items). Depression scale scores range from 0 to 42 with higher scores representing greater depression severity. Anxiety scale scores range from 0 to 42 with higher scores representing greater anxiety severity. Stress scale scores range from 0 to 42 with higher scores representing greater stress.
Pregnancy-related Empowerment | 6 months
  Assess feelings of empowerment related to pregnancy (via PRES, the Pregnancy-Related Empowerment Scale). Scores range from 16 to 64, with higher scores representing stronger feelings of pregnancy-related empowerment.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No